CLINICAL TRIAL: NCT04769986
Title: Development of a Mobile Mindfulness Intervention for Alcohol Use Disorder and PTSD Among OEF/OIF Veterans
Brief Title: Mobile Mindfulness for Alcohol Use and PTSD Among Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); National Center for PTSD (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Pedersen, Associate Professor of Psychiatry and the Behavioral Sciences and Population and Public Health Sciences, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34AA027845-01 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-25 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Use Disorder; Posttraumatic Stress Disorder
Keywords: Veterans; Mindfulness; Alcohol
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Mindfulness-Based Relapse Prevention (mMBRP) (Experimental): Participants will complete the Mindfulness Coach app program that is enhanced with additional modules containing MBRP content.
  Interventions: Behavioral: Mobile Mindfulness-Relapse Prevention (mMBRP)
- Active control (Active Comparator): Participants will complete a course of an exercise/healthy eating app program that is matched in time and effort to the intervention condition app.
  Interventions: Behavioral: Exercise/healthy eating mobile app

INTERVENTIONS:
Behavioral: Mobile Mindfulness-Relapse Prevention (mMBRP) — Mindfulness Coach 2.0 is a mobile application designed by the VA's National Center for PTSD. The app provides: (a) psychoeducational topics related to mindfulness; (b) audio-guided mindfulness exercises; (c) self-assessment using the Five Facet Mindfulness Questionnaire (d) a journal to track mindfulness practice sessions; (e) goal setting and tracking; (f) personal, customizable reminders; and (g) immediate access to support and crisis resources. We will enhance Mindfulness Coach with MBRP content by adding information about the triangle of awareness to understand connections among thoughts, sensations, and emotions, and specific meditations of sober breathing space and urge surfing to deal with cravings. We will add additional MBRP-specific modules. Participants will be asked to complete the intervention during 8 weeks, with two to three modules per week. After a beta test with 20 veterans, feedback will be used to refine the app for the national randomized clinical trial (RCT).
  Arms: Mobile Mindfulness-Based Relapse Prevention (mMBRP)
Behavioral: Exercise/healthy eating mobile app — Participants in the control condition will be asked to download an exercise/healthy eating mobile app and use it for 8 weeks. Similar to Mindfulness Coach, the app will have specialized self-management guides that follow a guide-per-week format, educational videos that teach diet and exercise strategies, and a diary to track diet and exercise progress.
  Arms: Active control

SUMMARY:
The purpose of the present study is to develop and test a mobile mindfulness intervention for Alcohol Use Disorder and PTSD among OEF/OIF veterans

DETAILED DESCRIPTION:
The long-term goal of this proposal is to improve treatment outcomes for OEF/OIF(Operation Enduring Freedom/Operation Iraqi Freedom) veterans with alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) who are not currently accessing care through the Veterans Affairs Healthcare System (VA) or other settings. Many OEF/OIF veterans struggle with heavy drinking and related consequences and this can be especially pronounced with the co-occurrence of PTSD. Prior research has found aspects of self-regulation (emotion regulation, impulse control), stress, and craving to be important putative targets in AUD and PTSD symptom reduction. However, with upwards of 50% of veterans who have behavioral health needs not seeking treatment, it is imperative to utilize advances in technology to develop and test interventions that can reach non-treatment seeking veterans and target both symptoms of PTSD and AUD. As the proposed mechanisms (e.g., self-regulation) are becoming better understood regarding how they affect PTSD and AUD outcomes, approaches should focus on targeting these mechanisms and evaluating if they are essential facilitators of change. Mindfulness-based interventions (MBI) can target such mechanisms, but a gap in the knowledge persists regarding the utility of MBIs with veterans who screen positive for PTSD and AUD. Therefore, we propose to improve treatment outcomes for OEF/OIF veterans with PTSD and AUD by targeting self-regulation, stress, and cravings. We will develop and test a novel mobile MBI, Mobile Mindfulness Based Relapse Prevention (mMBRP), that will improve upon evidence based in-person and group MBRP by reaching veterans outside of treatment settings. The engaging and easy to use mobile MBI integrates relapse prevention, stress reduction, and self-regulation skills and is relevant to issues surrounding stigma and barriers that veterans face when seeking services. The central hypothesis will be tested through a focus on three specific aims: (1) refine and add MBRP content to the popular VA developed Mindfulness Coach mobile application through a beta testing phase where we test for feasibility and acceptability of the app, (2) pilot test the efficacy of the mMBRP mobile app on alcohol use and PTSD outcomes compared to control, and (3) assess mechanisms of change such as self-regulation, stress, and cravings, as well as exploratory moderators of gender, race/ethnicity, and recency of discharge, on mMBRP effects. The unique strengths of this proposal are its focus on an underserved population, utilization of mobile technology for intervention delivery, and use of a novel intervention known to effectively target self-regulation and stress. The expected results will define a viable and easy-to-access treatment that can improve both AUD and PTSD symptoms. Results of this study will have a positive impact on substance use outcomes for those who have experienced traumatic events and will identify mechanism of action for treatment success. The app can be disseminated through our partners in the VA and through targeted sharing on social media.

ELIGIBILITY:
Inclusion Criteria:

* veterans aged 18 or older who have separated/discharged from military service from the Air Force, Army, Marine Corps, or Navy;
* have served as part of Operations Enduring Freedom, Iraqi Freedom, or New Dawn (OEF/OIF/OND)
* be able to read English
* own a personal smartphone with Internet access and be interested in using apps on that phone
* score 8 or higher on the Alcohol Use Disorder Identification Test, which represents probable AUD in civilian and military samples and is the VA's criteria for "severe risk" of AUD warranting referral to a substance use treatment clinic
* score a 33 or higher on the PTSD check list (PCL-5), which represents probable PTSD diagnosis among OEF/OIF veterans.

Exclusion Criteria:

* currently affiliated with active duty service or in the reserves or guard units
* past six-month treatment for alcohol or drug use or PTSD at the Veterans Affairs Healthcare System (VA) or other health care providers or clinics;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
change in PTSD symptoms | Time 1: baseline; Time 2: 4 week; Time 3: 8 week; Time 4: 12 week; Time 5: 16 week
  The PTSD Checklist is a 20-item self-report measure that assesses the 20 DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) symptoms of PTSD.
change in Alcohol use and related problems | Time 1: baseline; Time 2: 4 week; Time 3: 8 week; Time 4: 12 week; Time 5: 16 week
  Alcohol use will be measured using an online version of the timeline follow back, which will assess past 30 day drinking days and typical drinks per occasion. Number of alcohol consequences experienced in the past month will be assessed with the 24-item Brief Young Adult Alcohol Consequences Questionnaire.

SECONDARY OUTCOMES:
change in Treatment engagement | Screening in beta test; Time 1: baseline; Time 2: 4 week; Time 3: 8 week
  The Mental Health/Substance Use Disorder Treatment History Inventory will be used to screen in participants who have not used care in the past 6-months as well as examine if participants engage in care during the treatment phase or during the post-treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan P Davis, PhD, Principal Investigator — RAND; Eric R Pedersen, PhD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - National Center for PTSD, Menlo Park, California
  - San Francisco Veterans Affairs Healthcare System, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis JP, Pedersen ER, Borsari B, Bowen S, Owen J, Sedano A, Fitzke R, Delacruz J, Tran DD, Buch K, Saba S, Canning L, Bunyi J. Development of a mobile mindfulness smartphone app for post-traumatic stress disorder and alcohol use problems for veterans: Beta test results and study protocol for a pilot randomized controlled trial. Contemp Clin Trials. 2023 Jun;129:107181. doi: 10.1016/j.cct.2023.107181. Epub 2023 Apr 12. PMID 37059261